CLINICAL TRIAL: NCT03623464
Title: Randomized Clinical Trial of FitBit and Mobile Apps Versus Usual Care to Improve Post-Operative Outcomes After GI Cancer Surgery
Brief Title: RCT of Mobile Apps & FitBit v. Usual Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Damon Runyon Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1608017482
Record Dates: First submitted 2017-04-24; First posted 2018-08-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Cancer; Gastric Cancer; Hepatic Cancer; Colon Cancer; Rectal Cancer; Small Bowel Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms; Liver Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile app and Fitbit + Standard of care (Active Comparator): Mobile health application and Fitbit + standard of care: Participants will utilize mobile app and Fitbit and standard of care. Mobility data will be generated using a mobile health tracker designed for smartphone devices.
  Interventions: Other: Mobile health application and Fitbit + standard of care
- Standard of care (Other): Participants will receive standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Mobile health application and Fitbit + standard of care — Mobility data will be generated using a mobile health tracker designed for smartphone devices, which allows the phone to automatically and passively (no patient input needed) capture information on the patient's activity; i.e. if the person is walking, remaining stationary, or moving at a rapid speed (eg. in a car). The app will prompt patients once daily to answer a series of questions that will collect patient reported symptoms and health status data. Physicians will be alerted to abnormal values within 24-48 hours and patients will be triggered to call their physicians immediately if the values are outside of normal parameters.
  Arms: Mobile app and Fitbit + Standard of care
Other: Standard of care — Post-operative standard of care information
  Arms: Standard of care

SUMMARY:
This is a randomized clinical trial to evaluate the use of mobile devices in preventing readmission in patients undergoing major GI cancer operations.

DETAILED DESCRIPTION:
Patients will be randomized to 1) standard of care or 2) to use our mobile app with standard care. The mobile app will collect information on patients' daily physical activity patterns and health status data for clinicians using smartphone mobile technology applications. The investigators believe that by tracking information on patients, the investigators may be able to intervene sooner and prevent a delay in care.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subject speaks English
3. Subject owns a smart phone
4. Subject is scheduled to undergo surgery for a GI cancer (pancreatic, hepatic, gastric, small bowel, colon, or rectal cancers)

Exclusion Criteria:

1. Physician deems the subject is unable to complete the study due to documented dementia
2. Subject is undergoing emergent surgery
3. Subject has sepsis from another source
4. Physician deems the subject is unable to complete the study due to documented alcohol and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Readmission rate | 30 days
  Investigators will track readmission rates after surgery for those on the trial

SECONDARY OUTCOMES:
Healthcare utilization rates | 30 days
  Investigators will track patients' healthcare resource utilization and the cost of this utilization by assessing how often the patients contact their providers via phone or the app, access the emergency room, and through readmission data.
Patient Satisfaction with Device | 30 days
  Investigators will assess patients' satisfaction with their care experience and device. This will be done with an internal questionnaire asking if patients were satisfied and if they found it easy to use.
Quality of life: Return to Baseline Function-Walking | 30 days
  Investigators will monitor patients' return to baseline health after surgery by tracking progress via step counts, as monitored by a FitBit tracker.
Quality of life: Return to Baseline Function-Activities of Daily Living (ADLs) | 30 days
  Investigators will monitor patients' return to baseline health after surgery by tracking progress using a questionnaire, modified from the Katz Activities of Daily Living scale. For this scale, a score of 6 is high, indicating that the patient is independent and a score of 0 is low, indicating that the patient very dependent in performing their ADLs.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Yeo, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine- New York Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No